CLINICAL TRIAL: NCT01065064
Title: Visual Performance After Implantation of an Aspheric Multifocal Diffractive Intraocular Lens
Brief Title: Visual Performance After RESTOR Implantation
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hospital Oftalmologico de Brasilia (Other)
Responsible Party: PATRICK FRENSEL DE MORAES TZELIKIS, HOSPITAL OFTALMOLOGICO DE BRASILIA; UFMG; HBDF
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: HOB-01/09
Record Dates: First submitted 2010-02-08; First posted 2010-02-09 (Estimated); Last update posted 2010-02-09 (Estimated); Status verified 2010-02

CONDITIONS: Refractive Assessment
Keywords: Multifocal IOL; ReSTOR IOL

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- RESTOR (Experimental): Patients with cataract that had phacoemulsification and AcrySof® ReSTOR IOL implantation.
  Interventions: Procedure: RESTOR IOL

INTERVENTIONS:
Procedure: RESTOR IOL — The U.S. Food and Drug Administration (FDA) has granted approval of Alcon's AcrySof® ReSTOR® intraocular lens (IOL) for cataract patients with and without presbyopia. This innovative lens uses a revolutionary apodized diffractive technology to give patients a full range of quality vision (near, intermediate and distance) that greatly increases their independence from glasses after surgery
  Other Names: RESTOR IQ MULTIFOCAL IOL

SUMMARY:
The purpose of this study is to evaluate the distance, intermediate, and near vision after aspheric multifocal diffractive AcrySof® ReSTOR SN6AD1 intraocular lens (IOL) implantation.

DETAILED DESCRIPTION:
To evaluate distance, intermediate, and near vision after aspheric multifocal diffractive AcrySof® ReSTOR SN6AD1 intraocular lens (IOL) implantation.

Prospective study of 50 patients with cataract that had phacoemulsification and AcrySof® ReSTOR IOL implantation. Uncorrected distance vision acuity (UDVA), corrected distance visual acuity (CDVA), distance-corrected near visual acuity (DCNVA), and distance-corrected intermediate visual acuity (DCIVA) were measured postoperatively. A patient-satisfaction and visual phenomena questionnaire was administered at the end of the study.

ELIGIBILITY:
Inclusion Criteria:

* Cataract
* Any race
* Either gender
* Diagnosis of cataracts both eyes
* Pre-existing physical conditions that could skew visual results, such as Diabetes, Retinal detachment, Macular degeneration, or Cancer
* Subjects must have < 1.00 diopter of astigmatism
* Biometry results for the Restore patients should target emmetropia or +0.25.

Exclusion Criteria:

* Central endothelial cell count less than 2000 cells/mm2 glaucoma or intraocular pressure greater than 21 mmHg amblyopia
* Retinal abnormalities
* Diabetes mellitus steroid or immunosuppressive treatment
* Connective tissue diseases

Ages: 45 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2009-01; Primary Completion 2009-02 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
To evaluate distance, intermediate, and near vision after aspheric multifocal diffractive AcrySof® ReSTOR SN6AD1 intraocular lens (IOL) implantation. | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: PATRICK F TZELIKIS, MD, PhD, Principal Investigator — HOB; HBDF; UFMG
Locations (1):
- Hospital Oftalmologico de Brasilia, Brasília, Federal District, Brazil

REFERENCES:
- [Background] Artem'eva LS, Asin BA, Guliaev AA. [Method of prolonged active drainage after operations on the joints in rheumatoid arthritis]. Ortop Travmatol Protez. 1979 Aug;(8):28-9. No abstract available. Russian. PMID 503440
- [Result] Kohnen T, Nuijts R, Levy P, Haefliger E, Alfonso JF. Visual function after bilateral implantation of apodized diffractive aspheric multifocal intraocular lenses with a +3.0 D addition. J Cataract Refract Surg. 2009 Dec;35(12):2062-9. doi: 10.1016/j.jcrs.2009.08.013. PMID 19969209
- [Result] Alfonso JF, Fernandez-Vega L, Orti S, Ferrer-Blasco T, Montes-Mico R. Refractive and visual results after implantation of the AcrySof ReSTOR IOL in high and low hyperopic eyes. Eur J Ophthalmol. 2009 Sep-Oct;19(5):748-53. doi: 10.1177/112067210901900511. PMID 19787593